CLINICAL TRIAL: NCT06275932
Title: Management of Healthy Newborn's Body Temperature With the Use of Blanket: Randomized Controlled Trial
Brief Title: Management of Healthy Newborn's Body Temperature at Birth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TermoNeo/2023
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Newborn, Infant; Body Temperature; Delivery Room
Keywords: newborn, infant; body temperature; delivery room; hypothermia, induced
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): All the enrolled newborns will make the skin-to-skin contact with the use of a thermal blanket after birth.
  Interventions: Other: Interventional group
- Standard of care group (Active Comparator): All the enrolled newborns will make the skin-to-skin contact according to local procedure after birth.
  Interventions: Other: Standard of care group

INTERVENTIONS:
Other: Interventional group — Newborns will be covered with a thermal blanket during skin-to-skin contact in delivery room.
  Arms: Interventional group
Other: Standard of care group — Newborns will be covered with a bed wetting mat and cotton sheet during skin-to-skin contact in delivery room.
  Arms: Standard of care group

SUMMARY:
At birth, the newborn begins a process of adaptation to extrauterine life. One of the phases of this stabilization process is the maintenance of body temperature; indeed, the newborn passes from a warm environment (mother's womb) of around 37°C to an environment with a temperature lower (delivery room) and, therefore, must implement a series of physiological processes to be able to maintain body temperature constant and within ideal ranges through a balance between production and heat loss.

Hypothermia at birth could cause risks or comorbidities such as an increased risk of infant mortality, hypoglycemia, sepsis, metabolic acidosis, respiratory distress syndrome (RDS) and intraventricular hemorrhage (IVH).

One of the factors that affects heat loss in the delivery room is the relationship between surface area, volume and body mass of the newborn. The decrease in body temperature is directly related to gestational age and weight at birth; indeed, this problem is much more present in premature and/or low weight newborns at birth. Even if a full-term newborn has a more developed thermoregulation center than a preterm newborn, this does not mean that this type of newborns is not at risk heat dispersion.

To date, the strategies that are implemented for the physiological newborn are documented in the literature are, in addition to the heat chain described by the World Health Organization (WHO), the implementation of skin-to-skin contact (skin to skin) mother-newborn.

Some studies demonstrating the beneficial effect of this procedure on maintenance of the newborn's body temperature.

The aim of this study is to evaluate two healthcare interventions to prevent heat loss of healthy newborns at birth.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial design which involves the use of two care interventions (experimental vs standard of care) to prevent heat loss of healthy newborns in the delivery room during contact skin to skin after birth.

Study population includes newborns born by natural birth with a gestational age greater than or equal to 37+0 weeks.

Newborns will be randomly assigned to receive: 1) a thermal blanket (experimental group) , or 2) a bed wetting mat and cotton sheet (standard of care group) that cover them during the skin-to-skin contact after birth.

At birth all newborns will receive the same care required by local procedures.

Research hypothesis:

- the use of a thermal blanket placed on the newborn during the skin-to-skin contact could reduce heat dispersion at the end of the procedure and therefore reduce the percentage of newborns who at the end of skin-to-skin contact have a temperature lower than 36.5°C.

The effectiveness of these interventions will be evaluated by measuring mother and newborn's body temperature at the beginning and the end of skin-to-skin contact.

ELIGIBILITY:
Inclusion Criteria:

For mother

* Mothers' age over 18 years and good comprehension of Italian language;
* Signed informed consent of the mother.

For newborn

* Informed consent signed by both parents, or in the case of a single-parent family, by mother
* Gestational age at birth greater than or equal to 37+0 weeks
* Newborns from singleton pregnancies;
* Both male and female newborns;
* Newborns who will be born from vaginal birth.

Exclusion Criteria:

For mother

* Mothers who do not want to carry out skin-to-skin contact;
* Mothers who do not understand/speak the Italian language;
* Mothers who need assistance procedures that hinder skin-to-skin contact.

For newborn

* Newborns whose parents decline participation in the study;
* Newborns with major congenital anomalies (heart, brain, metabolic, gastrointestinal);
* Newborns born via cesarean section;
* Newborns whose parents are under 18 years old, in the case of a single parent the mother who is under 18 years;
* Newborns requiring neonatal resuscitation after birth with obstruction of the skin-to-skin contact.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 776 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Newborn's body temperature at the end of skin-to-skin contact | At the beginning and the end skin-to-skin contact, up to three hours after birth.
  Newborn's body temperature will be measured at the beginning and the end of skin-to-skin contact with a digital thermometer placed in axillary location. Newborn's body temperature at the end of kin-to-skin contact will be compared between two groups.

SECONDARY OUTCOMES:
Newborns' proportion with a body temperature < 36.5°C when arriving at the nursery | At the arrival in the nursery, up to six hours after birth.
  Evaluation of newborns' proportion with a body temperature < 36.5°C will be calculated in both arms of study measuring newborn's body temperature with a digital thermometer placed in axillary location when they will arrive at the nursery.
Newborns' proportion with temperature below 36.0°C at the end of skin-to-skin contact and at arrival in the nursery | At the end of skin-to-skin contact and at arrival in the nursery, up to six hours after birth.
  Evaluation of newborns' proportion with temperature below 36.0°C at the end of skin-to-skin contact and at arrival in the nursery, in variation of the time spent in the delivery room at the end of the skin-to-skin contact, will be calculated in both arms of study measuring newborn's body temperature with a digital thermometer placed in axillary location.
Newborns' proportion with moderate hypothermia (temperature 36.0 - 36.4°C) at the end of skin-to-skin contact and at arrival in the nursery | At the end of skin-to-skin contact and at arrival in the nursery, up to six hours after birth.
  Evaluation of newborns' proportion with moderate hypothermia (temperature 36.0 - 36.4°C) at the end of skin-to-skin contact and at arrival in the nursery, in variation of the time spent in the delivery room at the end of the skin-to-skin contact, will be calculated in both arms of study measuring newborn's body temperature with a digital thermometer placed in axillary location.
Newborns' proportion with hyperthermia (temperature > 37.5°C) at the end of skin-to-skin contact and at arrival in the nursery | At the end of skin-to-skin contact and at arrival in the nursery, up to six hours after birth.
  Evaluation of newborns' proportion with hyperthermia (temperature > 37.5°C) at the end of skin-to-skin contact and at arrival in the nursery, in variation of the time spent in the delivery room at the end of the skin-to-skin contact, will be calculated in both arms of study measuring newborn's body temperature with a digital thermometer placed in axillary location.
Newborns' average temperature one hour after arriving at the nursery | At arrival in the nursery, up to six hours after birth.
  Evaluation of newborns' average temperature one hour after arriving at the nursery will be calculated in both arms of study measuring newborn's body temperature with a digital thermometer placed in axillary location.
Duration of nursery stay | from birth until discharge, measured up to 1 week.
  Duration of stay in the nursery (hours) will be collected from electronical medical records
Duration of skin-to-skin contact | From the beginning until the end of skin-to-skin contact, up to three hours after birth.
  Duration of skin-to-skin contact (minutes) will be collected from electronical medical records
Newborns' proportion exclusively breastfed at discharge | At discharge from the nursery, measured up to 1 week.
  Evaluation of Newborns' proportion exclusively breastfed at discharge will be collected from electronical medical records
Type of breastfeeding at discharge | At discharge from the nursery, measured up to 1 week.
  Evaluation of the type of breastfeeding at discharge will be collected from electronical medical records.
Newborns' proportion with hypoglycemia during hospitalization | At discharge from the nursery, measured up to 1 week.
  Evaluation of newborns' proportion with hypoglycemia during hospitalization will be collected from electronical medical records
Newborns' proportion affected by respiratory distress syndrome | At discharge from the nursery, measured up to 1 week.
  Evaluation of newborns' proportion affected by respiratory distress syndrome will be collected from electronical medical records.
Newborns' proportion transferred to the Neonatal Intensive Care Unit (NICU) | At discharge from the nursery, measured up to 1 week.
  Evaluation of newborns' proportion transferred to the NICU will be collected from electronical medical records.
Newborns' weight loss at discharge | At discharge from the nursery, measured up to 1 week.
  Percentage of Newborns' weight loss at discharge will be collected from electronical medical records.
Mortality before discharge from hospital | At discharge from the nursery, measured up to 1 week.
  Evaluation of mortality before discharge from hospital will be collected from electronical medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Sorrentino, pedRN, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma D. Golden hour of neonatal life: Need of the hour. Matern Health Neonatol Perinatol. 2017 Sep 19;3:16. doi: 10.1186/s40748-017-0057-x. eCollection 2017. PMID 28932408
- [Background] Manani M, Jegatheesan P, DeSandre G, Song D, Showalter L, Govindaswami B. Elimination of admission hypothermia in preterm very low-birth-weight infants by standardization of delivery room management. Perm J. 2013 Summer;17(3):8-13. doi: 10.7812/TPP/12-130. PMID 24355884
- [Background] Trevisanuto D, Testoni D, de Almeida MFB. Maintaining normothermia: Why and how? Semin Fetal Neonatal Med. 2018 Oct;23(5):333-339. doi: 10.1016/j.siny.2018.03.009. Epub 2018 Mar 21. PMID 29599071
- [Background] World Health Organization. Thermal protection of the newborn: a practical guide. Published online 1997.
- [Background] Duryea EL, Nelson DB, Wyckoff MH, Grant EN, Tao W, Sadana N, Chalak LF, McIntire DD, Leveno KJ. The impact of ambient operating room temperature on neonatal and maternal hypothermia and associated morbidities: a randomized controlled trial. Am J Obstet Gynecol. 2016 Apr;214(4):505.e1-505.e7. doi: 10.1016/j.ajog.2016.01.190. Epub 2016 Feb 10. PMID 26874298
- [Background] Moore ER, Anderson GC, Bergman N, Dowswell T. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2012 May 16;5(5):CD003519. doi: 10.1002/14651858.CD003519.pub3. PMID 22592691
- See also: WHO Recommendations on Postnatal Care of the Mother and Newborn. World Health Organization — http://www.ncbi.nlm.nih.gov/books/NBK190086/